CLINICAL TRIAL: NCT06880939
Title: Randomized, Double-Blind, Parallel-Controlled, Multicenter Clinical Study on the Efficacy of Antarctic Krill Oil Functional Food in Alleviating Side Effects of Intravesical Therapy for Bladder Cancer
Brief Title: Antarctic Krill Oil Functional Food Mitigates Bladder Cancer Treatment Side Effects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYLL-202412-011-1
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Bladder Cancer; Krill Oil; Intravesical Therapy; Adverse Effects; Randomized Controlled Trial
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: 1. Experimental Group:
     Dosage: Oral administration of 2g krill oil daily. The krill oil supplement is provided in 1g capsules, with one capsule taken 30 minutes after breakfast and one capsule 30 minutes after dinner.
     Duration: The supplementation begins on the day of the first bladder instillation treatment and continues until the day of the last bladder instillation treatment.
  2. Control Group:
  Intervention: No krill oil is administered. Instead, a placebo capsule with a similar appearance is used, containing olive oil. The placebo is provided in 1g capsules, with one capsule taken 30 minutes after breakfast and one capsule 30 minutes after dinner.
  Duration: The placebo administration begins on the day of the first bladder instillation treatment and continues until the day of the last bladder instillation treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the participants and investigators are unaware of the group assignments, and the entire trial is arranged and controlled by the study designer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Krill Oil Functional Food Group (Experimental): Dosage: 2 g of krill oil per day, orally administered. Specification: Krill oil capsules are provided in 1 g/capsule format. Administration: Take 1 capsule 30 minutes after breakfast and 1 capsule 30 minutes after dinner.
  Note: The Antarctic krill oil functional food used in this study is produced and supplied by Jinan Jiyuan Biotechnology Co., Ltd. Its main components include phospholipids, DHA, EPA, and astaxanthin.
  Duration: Administration begins on the day of the first bladder instillation treatment and continues until the day of the last bladder instillation treatment.
  Form: Capsule form for convenient oral administration.
  Interventions: Dietary Supplement: Krill Oil Functional Food
- Olive Oil Group (Placebo Comparator): Intervention:Participants will not orally consume krill oil. Instead, they will receive placebo capsules that are visually identical to krill oil capsules.The placebo capsules contain olive oil.Each capsule is 1g in size.
  Dosage and Administration:Take 1 capsule after breakfast and 1 capsule after dinner, within 30 minutes of each meal.
  Duration:The intervention will begin on the day of the first bladder instillation treatment.It will continue until the day of the last bladder instillation treatment.
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Krill Oil Functional Food — Take 2g of krill oil orally daily, with each krill oil capsule containing 1g, by consuming one capsule within 30 minutes after breakfast and one capsule within 30 minutes after dinner. The supplementation period begins on the day of the first bladder instillation treatment and continues until the day of the last bladder instillation treatment.
  Arms: Krill Oil Functional Food Group
Dietary Supplement: Olive Oil — Instead of taking krill oil orally, use placebo capsules that are visually similar, with the contents being olive oil, each capsule containing 1g. Take one capsule within 30 minutes after breakfast and one capsule within 30 minutes after dinner. The duration of intake begins on the day of the first bladder instillation treatment and continues until the day of the last bladder instillation treatment.
  Arms: Olive Oil Group

SUMMARY:
This randomized, double-blind, placebo-controlled, multicenter trial evaluates the efficacy and safety of Antarctic krill oil in reducing side effects of intravesical therapy for non-muscle-invasive bladder cancer (NMIBC). A total of 210 participants (18-75 years) will be randomized to receive either 2g/day of krill oil capsules (containing phospholipids, DHA, EPA, and astaxanthin) or placebo during intravesical treatment (epirubicin, pirarubicin, or BCG).

Primary outcomes include bladder irritation symptoms (IPSS score), systemic adverse events, hematuria, and urinary tract infections. Secondary outcomes assess quality of life (QoL). Safety will monitor adverse events per CTCAE v5.0.

The study follows GCP standards and includes rigorous data management and ethical oversight. Results may offer a dietary intervention to improve treatment tolerance and QoL for bladder cancer patients.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multicenter clinical trial aims to evaluate the efficacy and safety of Antarctic krill oil functional food in alleviating side effects of intravesical therapy for bladder cancer. The study will enroll 210 participants (105 per group) aged 18-75 years with histologically confirmed non-muscle-invasive bladder cancer (NMIBC) who are scheduled to undergo postoperative intravesical therapy (e.g., epirubicin, pirarubicin, or BCG). Participants will be randomized to receive either 2g/day of krill oil capsules (containing phospholipids, DHA, EPA, and astaxanthin) or placebo (olive oil capsules) during their intravesical treatment period.

The primary outcomes include the reduction in bladder irritation symptoms (assessed via IPSS score), incidence of systemic adverse events (e.g., nausea, fatigue), hematuria, and urinary tract infections. Secondary outcomes focus on quality of life (QoL) improvements using standardized questionnaires. Safety monitoring will track adverse events related to krill oil or intravesical therapy, graded per CTCAE v5.0 criteria.

Statistical analyses will compare groups using t-tests, chi-square tests, repeated-measures ANOVA, and Cox regression models. The study anticipates a medium effect size (d=0.5) with 90% power and accounts for a 20% dropout rate. Conducted across three centers in China (Qilu Hospital of Shandong University, Qingdao University Affiliated Hospital, and Shandong Provincial Hospital), the trial adheres to GCP standards and includes rigorous data management, adverse event reporting, and ethical oversight. Results may offer a novel dietary intervention to improve tolerance and quality of life for bladder cancer patients undergoing intravesical therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed bladder cancer: The patient needs to be diagnosed with bladder cancer through pathological examination and have undergone bladder cancer surgery.
* 2. Planned to receive bladder infusion therapy: Patients need to plan to receive bladder infusion therapy after surgery and agree to participate in the study.
* 3. Age range: 18 to 75 years old.
* 4. Normal blood, liver and kidney function: Laboratory tests showed that the patient's blood routine, liver function and kidney function were within the normal range.
* 5. Signed informed consent: The patient understands the content of the study and voluntarily signs the informed consent.

Exclusion Criteria:

* 1. Serious comorbidities: including but not limited to heart disease, severe liver and kidney insufficiency, uncontrolled hypertension, diabetes, etc.
* 2. History of allergies: Patients with a known history of allergy to krill oil or perfusion drug components.
* 3. History of prior chemotherapy: Patients who have received perfusion therapy prior to this study.
* 4. History of other malignant tumors: Patients with a history of other malignant tumors.
* 5. Pregnancy or lactation: Female patients who are pregnant or lactating.
* 6. Psychiatric illness: Patients with a history of severe psychiatric illness or currently receiving treatment for psychiatric illness.
* 7. Poor study compliance: Patients who believe that they are unable to complete the entire trial process as required by the study.
* 8. Other: Other conditions that the investigator considers unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
The degree of relief from bladder irritation symptoms. | From the start to the end of bladder instillation therapy，Monthly follow-up visits are continued until the end of perfusion therapy and last approximately 1 year
  To evaluate whether krill oil can significantly alleviate symptoms such as urgency, frequency, and pain during urination, a symptom scoring system (e.g., the International Prostate Symptom Score, IPSS) can be used
Incidence of systemic adverse reactions | From the start to the end of bladder instillation therapy，Monthly follow-up visits are continued until the end of perfusion therapy and last approximately 1 year
  Record and compare the systemic adverse reactions (such as nausea, fatigue, fever, rash, etc.) between the experimental group and the control group during the treatment period and after the treatment has concluded.
Incidence of Hematuria | From the start to the end of bladder instillation therapy，Monthly follow-up visits are continued until the end of perfusion therapy and last approximately 1 year
  Record and compare the occurrence of hematuria in the experimental group and the control group during and after treatment.
Incidence of urinary tract infection | From the start to the end of bladder instillation therapy，Monthly follow-up visits are continued until the end of perfusion therapy and last approximately 1 year
  Assess the frequency of urinary tract infections through routine urinalysis, urine culture, and symptom monitoring.

SECONDARY OUTCOMES:
Quality of life score | From the start to the end of bladder instillation therapy，Monthly follow-up visits are continued until the end of perfusion therapy and last approximately 1 year
  The quality of life of study participants during and after treatment was assessed using the Quality of Life Scale (Qol) The quality of life of study participants during and after treatment was assessed using the Quality of Life Scale (Qol).

CONTACTS AND LOCATIONS:
Overall Officials: weiqiang Jing, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No